CLINICAL TRIAL: NCT04172116
Title: Continuous Glucose Monitoring (CGM) After Surgical Variations of the Roux-en-y Gastric Bypass: Comparing Tissue Glucose Levels Between Two Surgical Bypass Methods - a Prospective Study
Brief Title: Continuous Glucose Monitoring (CGM) After Surgical Variations of the Roux-en-y Gastric Bypass
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Gerhard Prager, Univ.Doz.Prof. Dr., Medical University of Vienna
Other Study IDs: 2235/2018
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Continuous Glucose Monitoring; Roux-en-y Gastric Bypass; Hypoglycemia
Keywords: metabolic surgery
MeSH Terms: conditions — Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood chemistry testing for blood glucose levels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- long pouch RYGB: Patients with the variation of a long and narrow pouch (hypothesis: slower transit of food)
  Interventions: Device: Continuous glucose monitoring
- short pouch RYGB: Patients with the variation of a short and wide pouch (hypothesis: faster pouch emptying as compared with long and narrow pouch)
  Interventions: Device: Continuous glucose monitoring

INTERVENTIONS:
Device: Continuous glucose monitoring — see arm/group descriptions

SUMMARY:
This study evaluates the difference in post prandial tissue glucose levels between two variation of Roux-en-Y Gastric bypass by continuous glucose monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent bariatric-metabolic surgery at the Medical University of Vienna in the years 2012-2016 for the "long and narrow" pouch group
2. Patients who underwent bariatric-metabolic surgery at the Clinic of Hollabrunn in the years 2010- 2012 for the "short and wide" pouch group
3. Patients on oral medication for diabetes mellitus (for subgroup assessment)
4. Stable weight (not more than + 15kg from lowest weight postoperatively)
5. Stable BMI

Exclusion Criteria:

1. Unable to give written informed consent
2. Patients with methods other than RYGB
3. Reoperation within the observed period
4. Any intervention changing pouch size or diameter of the anastomosis after the initial operation
5. Known allergy to oral contrast agent
6. Any regular intake of medication interfering with blood glucose levels

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Of each bariatric-metabolic operation we plan to include 34 patients. Of these 34 patients we plan to include also patients in each group with a diagnosed Diabetes mellitus type II at the time of operation (defined by either HbA1c >6.5 or any medication or impaired fasting blood glucose level)
  1. Roux-en-y gastric bypass with long ang narrow pouch ("long pouch RYGB")
  2. Roux-en-y gastric bypass with short and broad pouch ("short pouch RYGB")
  Patients in the two RYGB groups will be matched for sex, age, comorbidities and BMI at the time of operation.
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Tissue glucose levels | 6 days
  Difference in tissue glucose levels after the two variations of the Roux-en-y Gastric bypass

SECONDARY OUTCOMES:
tissue vs. blood glucose levels | 1 day
  Comparison of tissue and blood glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Prager, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Landesklinikum Weinviertel Hollabrunn, Hollabrunn, Austria

IPD SHARING:
Plan to Share IPD: No